CLINICAL TRIAL: NCT00425451
Title: The Efficacy and Safety of PerioChip Plus (Flurbiprofen/Chlorhexidine) Formulation in the Therapy of Adult Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dexcel Pharma Technologies Ltd. (Industry)
Responsible Party: Dr. Avi Avramoof/ V.P R&D, Dexcel Pharma Technologies Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLI/006P
Record Dates: First submitted 2007-01-21; First posted 2007-01-23 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Periodontitis
Keywords: Periodontitis; Dental Care; Efficacy; Safety
MeSH Terms: conditions — Periodontitis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- PerioChip Plus (Experimental)
  Interventions: Drug: PerioChip Plus (Flurbiprofen +Chlorhexidine ), Flurbiprofen Chip, PerioChip (Chlorhexidine ) and Placebo Chip
- Flurbiprofen Chip (Experimental)
  Interventions: Drug: PerioChip Plus (Flurbiprofen +Chlorhexidine ), Flurbiprofen Chip, PerioChip (Chlorhexidine ) and Placebo Chip
- PerioChip (Active Comparator)
  Interventions: Drug: PerioChip Plus (Flurbiprofen +Chlorhexidine ), Flurbiprofen Chip, PerioChip (Chlorhexidine ) and Placebo Chip
- Placebo Chip (Placebo Comparator)
  Interventions: Drug: PerioChip Plus (Flurbiprofen +Chlorhexidine ), Flurbiprofen Chip, PerioChip (Chlorhexidine ) and Placebo Chip

INTERVENTIONS:
Drug: PerioChip Plus (Flurbiprofen +Chlorhexidine ), Flurbiprofen Chip, PerioChip (Chlorhexidine ) and Placebo Chip

SUMMARY:
The purpose of this study is to determine the effect of the placement of a PerioChip Plus (flurbiprofen/chlorhexidine - FBP/CHX) formulation versus PerioChip (chlorhexidine) formulation versus Flurbiprofen Chip formulation versus Placebo Chip formulation on probing pocket depth (PPD)

DETAILED DESCRIPTION:
This is an 80 subjects, single-center, randomized, double-blinded, parallel, 4-arm clinical study (25 subjects in the PerioChip Plus and PerioChip arms and 15 subjects in the Flurbiprofen Chip and Placebo Chip arms).

At 24 weeks, relative to baseline, the mean reductions in probing pocket depth (PPD) will be used as primary efficacy endpoint. Additional primary endpoints are clinical attachment levels (CAL) and bleeding on probing (BOP) in the target pockets selected at screening, measured at weeks 24.

PPD measurements at 6, 12 and 18 weeks will be used as secondary endpoints. Additional secondary endpoints are clinical attachment levels (CAL) and bleeding on probing (BOP) in the target pockets selected at screening, measured at weeks 6, 12 and 18.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Good general health
* Male or female subjects aged >25 years old
* Minimum of 8 natural teeth
* Availability for the 25 weeks duration of the study
* Periodontal disease on a natural teeth characterized by the presence of at least 2 teeth with periodontal pockets of 6-9 mm in depth (target teeth) in order to reach baseline (day 1) with periodontal pockets of 5-8 mm in depth, without involving the apex of the tooth.
* Females of childbearing potential must be non pregnant at entry and agree to use an adequate method of birth control during the study.
* Demonstrate bleeding on probing to the base of the pocket at the pockets (sites) selected at the time of screening.

Exclusion Criteria:

* Presence of oral local mechanical factors that could (in the opinion of the investigator) influences the outcome of the study.
* Presence of orthodontic appliances or any removable appliance that impinges on the tissues being assessed.
* Soft or hard tissue tumours of the oral cavity.
* Presence of dental implant adjacent to target tooth.
* Periodontal pockets of more than 9 mm in depth.
* General systemic antibiotics therapy or periodontal/mechanical/local delivery therapy within 6 weeks prior to study entry and through out the study duration.
* History of allergy to chlorhexidine, flurbiprofen or to other non-steroidal anti-inflammatory drugs (NSAIDs).
* Subjects taking diphenylhydantoin, nifedepine and/or cyclosporine, which might influence the pattern of tissue response.
* Subject treated with non-steroidal anti-inflammatory drugs (NSAIDs) within 14 days prior to entry into the study and through out the study duration.
* Pregnant women or those planning to become pregnant or lactating women.
* Presence of the following conditions: Type 1 diabetes, major recurrent aphtae, stomatitis and related oral pathologies.
* The presence of any medical or psychiatric condition or any other condition that in the opinion of the investigator could affect the successful participation of the subject in the study.
* Subject participates in any other clinical study 30 days prior to the start of the study and through out the study duration.
* Subject uses chlorhexidine oral rinses/ mouthwashes on a regular basis.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
At 24 weeks, relative to baseline, the mean reductions in probing pocket depth (PPD) will be used as primary efficacy endpoint. Additional primary endpoints are clinical attachment levels (CAL) and bleeding on probing (BOP) in the target pockets selected | 24 weeks

SECONDARY OUTCOMES:
PPD measurements at 6, 12 and 18 weeks will be used as secondary endpoints. Additional secondary endpoints are clinical attachment levels (CAL) and bleeding on probing (BOP) in the target pockets selected at screening, measured at weeks 6, 12 and 18. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aubrey Soskolne, Professor, Principal Investigator — Hadassah Medical Organization IRB
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel